CLINICAL TRIAL: NCT01794351
Title: Effects of Trans-resveratrol on Cognitive Performance in Healthy, Young Humans: a Double-blind, Placebo-controlled, Crossover Investigation.
Brief Title: Cognitive Effects of 500mg Trans-resveratrol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, David Kennedy, Professor, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 22P5
Record Dates: First submitted 2013-02-08; First posted 2013-02-18 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Cognitive Performance; Mood
MeSH Terms: interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo then resveratrol (Experimental): Participants in this arm (decided according to Latin square) first received placebo and then resveratrol, on seperate days, with a 7-14 day wash-out period between visits.
  Interventions: Dietary Supplement: Trans-resveratrol; Other: Placebo
- Resveratrol then placebo (Experimental): Participants in this arm (decided according to Latin square) first received resveratrol and then placebo, on seperate days, with a 7-14 day wash-out period between visits
  Interventions: Dietary Supplement: Trans-resveratrol; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Trans-resveratrol — In this crossoevr study, all participants also consumed 500mg trans-resveratrol (in 2 opaque vegetarian capsules), at baseline, on counterballanced days.
Other: Placebo — In this crossoevr study, all participants also consumed placebo (2 opaque vegetarian capsules), at baseline, on counterballanced days.
  Other Names: Pharmaceutical grade silica

SUMMARY:
This study investigated the potentially cognitive enhancing effects of 500mg trans-resveratrol in healthy, young humans.

ELIGIBILITY:
Inclusion Criteria:

* 18-35yrs, healthy.

Exclusion Criteria:

* Drug/alcohol abuse, taking prescription medication (apart from contraception) or herbal supplements, having food intolerances or allergies, having suffered a head-injury or neurological/neuro-developmental disorder, uncorrected sight problems, pregnant or seeking to become so, excessive caffeine use (e.g. more than 6 cups of coffee per day).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with altered cognitive function at 40mins post-dose | 40mins Post-dose
  This outcome measure is assessed by the number of participants whose scores on a range of cognitive tasks (word and picture recall and recognition, serial 3s and 7s subtractions, rapid visual information processing (RVIP), N-Back (3-Back version), Stroop and numeric working memory) differed from the baseline to 40min post-dose scores.
Number of participants with altered cognitive function at 2.5hrs post-dose | 2.5hrs post-dose
  This outcome measure is assessed by the number of participants whose scores on a range of cognitive tasks (word and picture recall and recognition, serial 3s and 7s subtractions, rapid visual information processing (RVIP), N-Back (3-Back version), Stroop and numeric working memory) differed from baseline to the 2.5hr post-dose scores.
Number of participants with altered cognitive function at 4hrs post-dose | 4hrs post-dose
  This outcome measure is assessed by the number of participants whose scores on a range of cognitive tasks (word and picture recall and recognition, serial 3s and 7s subtractions, rapid visual information processing (RVIP), N-Back (3-Back version), Stroop and numeric working memory) differed from baseline to the 4hr post-dose scores.
Number of participants with altered cognitive function at 6hrs post-dose | 6hrs post-dose
  This outcome measure is assessed by the number of participants whose scores on a range of cognitive tasks (word and picture recall and recognition, serial 3s and 7s subtractions, rapid visual information processing (RVIP), N-Back (3-Back version), Stroop and numeric working memory) differed from baseline to the 6hr post-dose scores.

SECONDARY OUTCOMES:
Number of participants with altered mood at 40mins post-dose. | 40mins post-dose
  This outcome was assessed by the number of participants whose baseline mood scores (as assessed by the Bond-Lader mood scale which categorises 'alert', 'content' and 'calm') differed from the 40mins post-dose scores.
Number of participants with altered mood at 2.5hrs post-dose | 2.5hrs post-dose
  This outcome was assessed by the number of participants whose baseline mood scores (as assessed by the Bond-Lader mood scale which categorises 'alert', 'content' and 'calm') differed from the 2.5hrs post-dose scores.
Number of participants with altered mood at 4hrs post-dose | 4hrs pos-dose
  This outcome was assessed by the number of participants whose baseline mood scores (as assessed by the Bond-Lader mood scale which categorises 'alert', 'content' and 'calm') differed from the 4hrs post-dose scores.
Number of participants with altered mood at 6hrs post-dose | 6hrs post-dose
  This outcome was assessed by the number of participants whose baseline mood scores (as assessed by the Bond-Lader mood scale which categorises 'alert', 'content' and 'calm') differed from the 6hrs post-dose scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Brain performance and nutrition research centre, Northumbria university, Newcastle upon Tyne, Tyne and Wear, United Kingdom